CLINICAL TRIAL: NCT01422421
Title: Intensive Blood Pressure and LDL Lowering for Better Survival and Cardiovascular Outcome in Diabetic Patients With Coronary Artery Disease: Randomized Controlled Trial
Brief Title: Intensive Blood Pressure and LDL Lowering in Diabetic Patients With Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeshi Morimoto (Other)
Collaborators: University of the Ryukyus (Other)
Responsible Party: Sponsor-Investigator, Takeshi Morimoto, Professor, Kyoto University, Graduate School of Medicine
Organization: Kyoto University, Graduate School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H21-rinsho shiken ippan-017
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease; Hypertension; Dyslipidemia
Keywords: type 2 diabetes; coronary artery disease; hypertension; dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Hypertension; Dyslipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intensive control (Active Comparator): systolic blood pressure less than 120mmHg and LDL cholesterol within 70- 85mg/dl
  Interventions: Other: intensive control
- standard control (Active Comparator): systolic blood pressure less than 130mmHg and LDL cholesterol less than 100mg/dl
  Interventions: Other: standard control

INTERVENTIONS:
Other: intensive control — use any medication to achieve systolic blood pressure less than 120mmHg and LDL cholesterol within 70-85mg/dl
  Arms: intensive control
Other: standard control — use any medication to achieve systolic blood pressure less than 130mmHg and LDL cholesterol less than 100mg/dl
  Arms: standard control

SUMMARY:
The purpose of this study is to determine whether intensive blood pressure and low density lipoprotein (LDL) cholesterol lowering could improve survival and cardiovascular outcome in Japanese diabetic patients with coronary artery disease and history of acute coronary syndrome.

DETAILED DESCRIPTION:
Prevalence of type 2 diabetes in Asia seems to be almost epidemic and establishment of preventive strategy against macrovascular as well as microvascular diseases are warranted because of higher cardiovascular risk in diabetic patients even without history of atherosclerotic cardiovascular diseases. Benefit of lowering low density lipoprotein (LDL) cholesterol down to 70 mg/ml in Caucasian patients with coronary artery disease (CAD) has been well established but not in Asian patients with lower risk of myocardial infarction and higher stroke risk. Intensive lowering blood pressure for cardiovascular outcome in diabetic patients and patients with CAD has been recommended in several guidelines without firm evidence. Risk and benefit of intensive blood pressure and LDL control should be evaluated in Japanese diabetic CAD patients by pragmatic randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with coronary artery disease and history of acute coronary syndrome
* Patients whose blood pressure and LDL cholesterol levels are above values recommended by the current guideline

Exclusion Criteria:

* Patients who have active malignant tumor
* Patients who are on hemodialysis due to end stage kidney disease
* Patients whom statins are contraindicated
* Patients who had acute coronary syndrome or stroke within 3 months
* Patients who are pregnant or on breast feeding
* Patients whose physicians deem that attending this trial is contraindicated or inappropriate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2011-08; Primary Completion 2022-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
composite endpoint | 3 years
  composite endpoint consisting of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke and unstable angina requiring hospital administration
important secondary composite endpoint | 3 years
  composite endpoint consisting of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke, unstable angina requiring hospital administration, and admission for heart failure

SECONDARY OUTCOMES:
all-cause mortality | 3 years
  death due to any cause
myocardial infarction | 3 years
  non fatal myocardial infarction
stroke | 3 years
  non fatal stroke excluding transient ischemic attack
Cardiovascular death | 3 years
  Cardiovascular death
end stage renal disease | 3 years
  end stage renal disease needs kidney transplantation or hemodialysis
peripheral artery disease | 3 years
  peripheral artery disease
new onset or deterioration of heart failure | 3 years
  new onset or deterioration of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Shinichiro Ueda, MD, PhD, Principal Investigator — Professor of Clinical Pharmacology and Therapeutics, University of the Ryukyus
Locations (2):
- Japan (2):
  - University Hospital, University of the Ryukyus, Nishihara, Okinawa
  - Saga University Hospital, Saga